CLINICAL TRIAL: NCT05874765
Title: A Study of Prevalence and Clinical Characteristics of Tic Disorders in Children at Sohag University Hospital
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Esraa Ahmed Mohamed, Resident-pediatric department-sohag hospital university, Sohag University
Other Study IDs: Soh-Med-23-04-19MS
Record Dates: First submitted 2023-05-16; First posted 2023-05-25 (Actual); Last update posted 2023-05-25 (Actual); Status verified 2023-05

CONDITIONS: Tic Disorder, Childhood
MeSH Terms: conditions — Tic Disorders | interventions — Diagnosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Diagnostic and Statistical Manual of mental disorder- fifth edition ( DSM5) — Diagnostic and Statistical Manual of mental disorder- fifth edition ( DSM5) , will be used to diagnose and classify the Tics among all included patients

SUMMARY:
Tics are brief, sudden, repetitive movements and/or sounds that increase with stress, anxiety, transitions, or excitement.

Tics occur most commonly in children and adolescents, with boys more frequently affected than girls The American Academy of Child and Adolescent Psychiatry states that tics affect up to 10 percent of children during their early school years. .

The exact pathophysiologic mechanisms are unknown, but the disorders are likely to be due to disturbances of the cortico striatal- thalamo -circuitry. Risk factors for tic disorders include. Genetics: Tics tend to run in families, so there may be a genetic basis to these disorders. Sex: Men are more likely to be affected by tic disorders than women.

They are divided into motor tics (e.g., blinking, shrugging shoulders, grimacing, or jerking) and vocal tics (e.g., throat clearing, sniffing, grunting) .

Patients describe an inner urge or a local premonitory sensation, which is then relieved by performing the tic. The tic can be voluntarily suppressed for short periods of time. Tics increase with stress, anxiety, transitions, and excitement, and decrease with distraction.

The American Academy of Child and Adolescent Psychiatry states that tics affect up to 10 percent of children during their early school years .The most notable tic disorder is Tourette syndrome, in which both physical and verbal tics occur in the same individual, often at the same time. Transient tic disorder also involves both types of tics, but they often occur individually .

Tic disorders are classified into 3 categories : Transient tic disorders involve motor or vocal tics that last for more than 4 weeks but less than a year. Chronic tic disorders involve either motor tics or vocal tics (but not both) that last for more than a year. Tourette Syndrome, in which both physical and verbal tics occur in the same individual Conditions associated with tic disorders, especially in children with TS, include: anxiety, ADHD, depression ,autism ,spectrum disorder learning difficulties ,OCD speech and language difficulties, sleep difficulties other complications associated with tic disorders are related to the effect of the tics on self-esteem and self-image . Some research! has found that children with TS or any chronic tic disorder experience a lower quality of life and lower self-esteem than those without one of these conditions

ELIGIBILITY:
Inclusion Criteria:

* -Age between 3 and 18 years
* All patients suffering from Tics and fulfill diagnostic criteria according to DSM V

Exclusion Criteria:

* - Patients with age below 3 years and after 18 years old

Ages: 3 Years to 18 Years | Sex: All
Age Groups: Child, Adult
Study Population: * -Age between 3 and 18 years
  * All patients suffering from Tics and fulfill diagnostic criteria according to DSM V
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-06 (Estimated); Primary Completion 2024-05 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Assessment of Tics severity will be by The Yale Global Tic Severity Scale ( Y G T S S-R) | 12 months
  A clinician-rated instrument considerd as the gold standard for assessing tics in patients with Trourettes Syndrome and other tic disorders

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag university Hospital, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Leckman JF, Riddle MA, Hardin MT, Ort SI, Swartz KL, Stevenson J, Cohen DJ. The Yale Global Tic Severity Scale: initial testing of a clinician-rated scale of tic severity. J Am Acad Child Adolesc Psychiatry. 1989 Jul;28(4):566-73. doi: 10.1097/00004583-198907000-00015. PMID 2768151
- [Background] Barker A, Musso MW, Jones GN, Roid G, Gouvier D. Unreliable block span reveals simulated intellectual disability on the stanford-binet intelligence scales-fifth edition. Appl Neuropsychol Adult. 2014;21(1):51-9. doi: 10.1080/09084282.2012.726670. Epub 2013 Jun 21. PMID 24826496